CLINICAL TRIAL: NCT07325669
Title: Comparison of the Effects of Total Intravenous Anaesthesia With Target-Controlled Infusion (TCI) and Inhalation Anaesthesia on Airway Complications During Extubation and in the Early Postoperative Period in Thyroidectomy Surgery
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: dilara gocmen (Other)
Responsible Party: Sponsor-Investigator, dilara gocmen, asst. Prof, Marmara University Pendik Training and Research Hospital
Organization: Marmara University Pendik Training and Research Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Screening
Other Study IDs: 2025/17/1234
Record Dates: First submitted 2025-12-11; First posted 2026-01-08 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2025-12

CONDITIONS: Throid Surgery; Airway Complication of Anaesthesia; Coughing Responses at Tracheal Extubation; Laryngospasm on Emergence; Target Controlled Infusion of Propofol; Sevoflurane Anaesthesia
Keywords: airway complication of anesthesia; tiroid surgery; propofol anesthesia

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group TIVA-TCI (Experimental): Anaesthesia induction will be achieved in all patients with 2 µg/kg remifentanil and 2-2.5 mg/kg propofol. In the TCI group, propofol will be administered using Medcaptain IV perfusors, with the target concentration at the site of action set at 3-4 µg/mL according to the Schneider model; remifentanil will be set at 2-4 ng/mL according to the Minto model (the CE certificate for the perfusor and TCI models is available and has been added to the file). All patients will receive rocuronium 0.6 mg/kg as a muscle relaxant, and intubation will be performed using an endotracheal tube with EMG electrodes. After intubation, the cuff pressure will be optimised to 20-30 cmH₂O using a manometer. No repeat muscle relaxant will be administered.
  During anaesthesia maintenance, propofol and remifentanil (propofol 3-4 µg/mL, remifentanil 2-4 ng/mL) will be administered via TCI in Group TIVA.
  Interventions: Drug: tıva
- Group Volatile anesthesia (Experimental): Anaesthesia induction will be achieved in all patients with 2 µg/kg remifentanil and 2-2.5 mg/kg propofol.
  In Group VA, sevoflurane MAC will be maintained at 1-1.2, and remifentanil infusion will be administered at a rate of 0.1-0.3 µg/kg/min.
  In both groups, anaesthesia depth will be monitored using BIS, and values will be maintained within the range of 40-60.
  Interventions: Drug: tıva

INTERVENTIONS:
Drug: tıva — In the TIVA group (total intravenous anaesthesia group), induction and maintenance of anaesthesia will be performed using target-controlled infusion (TCI) with propofol (Schneider model) and remifentanil (Minto model). In Group VA (volatile/inhalation anaesthesia group), maintenance anaesthesia will be administered with sevoflurane and remifentanil infusion following intravenous induction.
  Other Names: volatile agent

SUMMARY:
Thyroid surgery is one of the most complex operations in the head and neck region due to its close relationship with anatomical structures and the high risk of recurrent laryngeal nerve injury. The proximity of the surgical field to the trachea and larynx increases the likelihood of postoperative airway complications. Common complications include hypoparathyroidism (HP), recurrent laryngeal nerve (RLN) injury, injury to the external branch of the superior laryngeal nerve (EBLN), postoperative bleeding, thoracic canal injury, laryngeal oedema, tracheospasm, tracheal injury, and oesophageal injury. Serious complications such as dyspnoea, asphyxia, or thyroid crisis can lead to patient death.

Severe hypertension or coughing during awakening and extubation may cause bleeding from the surgical site, along with possible haematoma formation. In this context, safe extubation, maintenance of postoperative airway patency, and prevention of early complications are critical components of anaesthesia management in thyroid surgery.

Currently used anaesthesia techniques can directly affect the quality of the recovery process, the sensitivity of airway reflexes, and the reliability of nerve monitoring techniques. Total intravenous anaesthesia (TIVA) regimens, particularly when administered via target-controlled infusion (TCI) systems, allow for more precise control of anaesthetic depth and provide a more predictable, stable transition during the extubation period. In target-controlled intravenous anaesthesia, bolus and infusion of the anaesthetic agent are administered to achieve the desired target concentration based on the pharmacokinetic models of the drug according to the patient's age, gender, height, and weight. Various studies have indicated that the combination of propofol and remifentanil causes fewer complications such as agitation, coughing, and laryngospasm during the recovery period; in contrast, volatile agents such as sevoflurane may trigger undesirable effects such as increased secretion in the respiratory tract and laryngeal sensitivity more frequently.

Furthermore, intraoperative neuromonitoring (IONM) applications are increasingly being used to prevent recurrent laryngeal nerve injuries. However, the accuracy and signal quality of this technology are directly affected by the impact of the anaesthetic regimen on nerve-muscle transmission. The literature has shown that inhalation anaesthetics may weaken IONM responses by suppressing synaptic transmission, whereas TIVA provides more reliable and stable signal transmission. A study comparing propofol and inhalation anaesthesia in patients with papillary thyroid carcinoma showed that propofol-based total intravenous anaesthesia was associated with fewer postoperative recurrences.

In a study comparing TCI-TIVA and sevoflurane inhalation anaesthesia in laparoscopic cholecystectomy surgery, TCI was reported to be associated with less postoperative nausea and vomiting and haemodynamic instability. In a study involving 50 patients undergoing lumbar disc surgery who received general anaesthesia with sevoflurane-fentanyl and propofol-remifentanil, less coughing and haemodynamic instability during awakening were observed in the TIVA group.

The hypothesis of this study is that TIVA administered using the TCI method will result in fewer airway complications after extubation and higher intraoperative neuromonitoring signal quality compared to inhalation anaesthesia. The study will comparatively evaluate the advantages and disadvantages of two different anaesthesia techniques in terms of both postoperative airway safety and haemodynamics, as well as intraoperative nerve monitoring.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years or older,
* Classified as ASA I-II,
* Undergoing elective primary total or subtotal thyroidectomy surgery,
* Patients undergoing intraoperative neuromonitoring will be included in the study.

Exclusion Criteria:

* • History of difficult intubation,

  * History of neuromuscular disease,
  * Current vocal cord paralysis,
  * Previous neck surgery
  * Patients with a body mass index above 35 kg/m² were defined as morbidly obese.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2027-01-01 (Estimated); Study Completion 2027-03-01 (Estimated)

PRIMARY OUTCOMES:
postoperative cough score(0-3) | first 10 min after extubation
  Grade 0: No cough Grade 1: Mild, single cough Grade 2: Moderate cough lasting less than 5 seconds Grade 3: Severe, continuous cough lasting longer than 5 seconds (bucking)
postoperative laryngospasm score (0-3) | first 10 min after extubation
  Grade 0: No symptoms Grade 1: Stridor Grade 2: Complete obstruction of the vocal cords (breathing efforts without air movement) Grade 3: Cyanosis with evidence of airway obstruction at the level of the vocal cords.

SECONDARY OUTCOMES:
presence of post-extubation desaturation(spO2<92%) | first 30min after extubation
  An SpO2 level below 92% will be considered as indicating the development of postoperative desaturation.
requirement for re-intubation | first 30 min after extubation
  Re-intubation of a patient who cannot be ventilated or oxygenated after extubation
Positive pressure mask ventilation support | 30 min after extubation
  The need for chin lift and mask ventilation after extubation
postoperative care unit Richmond agitation scale score(+4,-5) | postoperative recovery period(30.min after extubation)
  postoperative care unit Richmond agitation scale score
  * 4 ->Combative-> Overtly combative or violent; immediate danger to staff
  * 3 ->Very agitated-> Pulls on or removes tube(s) or catheter(s) or has aggressive behavior toward staff
  * 2 Agitated ->Frequent nonpurposeful movement or patient-ventilator dys-synchrony
  * 1 Restless Anxious or apprehensive but movements not aggressive or vigorous 0 Alert and calm Spontaneously pays attention to caregiver
    * 1 Drowsy Not fully alert, but has sustained (more than 10 seconds) awakening, with eye contact, to voice
    * 2 Light sedation Briefly (less than 10 seconds) awakens with eye contact to voice
    * 3 Moderate sedation Any movement (but no eye contact) to voice
    * 4 Deep sedation No response to voice, but any movement to physical stimulation
    * 5 Unarousable No response to voice or physical stimulation

IPD SHARING:
Plan to Share IPD: Undecided